CLINICAL TRIAL: NCT01712776
Title: Prospective, Randomized, Blinded,Comparative Efficacy and Safety Trial of Vapocoolant (Pain Ease Medium Stream) for Venipuncture
Brief Title: Vapocoolant (Pain Ease) Use for Venipuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Gebauer Company (Network)
Responsible Party: Principal Investigator, Sharon Mace, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEB-01
Record Dates: First submitted 2012-10-04; First posted 2012-10-24 (Estimated); Results first posted 2014-12-11 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Pain
Keywords: Vapocoolant
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vapocoolant (Pain Ease Medium Stream ) (Active Comparator): Application of Vapocoolant (Pain Ease Medium Stream) for 4-10 seconds onto venipuncture site.
  Interventions: Device: Vapocoolant (Pain Ease)
- Nature's Tears Sterile Water (Placebo Comparator): Application of sterile water stream (nature's tears) for 4-10 seconds onto the venipuncture site.
  Interventions: Device: Nature's Tears Sterile Water

INTERVENTIONS:
Device: Vapocoolant (Pain Ease) — Topical stream 4-10 seconds duration to skin.
  Other Names: Pain Ease Stream
  Arms: Vapocoolant (Pain Ease Medium Stream )
Device: Nature's Tears Sterile Water — Topical stream 4-10 seconds duration to skin
  Arms: Nature's Tears Sterile Water

SUMMARY:
To determine the efficacy and safety of vapocoolant spray (Pain Ease Medium Stream) in decreasing the pain of venipuncture ("blood draw")

DETAILED DESCRIPTION:
This is a prospective, randomized, blinded, comparator study. This study design is considered standard for establishing safety and efficacy data. Active treatment vapocoolant spray (Pain Ease Medium Stream) spray) will be used. There will be a placebo (sterile water) in this study. The population selected for this study, adults (excluding the very old, > 80 years old) represents a patient population that may benefit from vapocoolant spray. This is a patient population that according to the treating health care provider already requires venipuncture for "blood draw" but not intravenous cannulation. Because venipuncture is a painful procedure, vapocoolant may confer benefit for the relief of pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient needing venipuncture ("blood draw') but not intravenous cannulation
* Adult 18 years and older up to and and including 80 years old
* Stable patient
* Mentally competent patient able to understand the consent form

Exclusion Criteria:

* Patients with any allergies to the spray components (e.g. 1,1,1,3,3 pentafluoropropane or 1,1,1,2, tetrafluoroethane )
* Critically ill or unstable (e.g. sepsis or shock)
* Extremes of age: geriatric (> 80 years) or pediatric ( < 18 years old)
* Pregnant
* Venipuncture site located in area of compromised blood supply. Examples include : patients with peripheral vascular disease, gangrene, Raynaud's disease, Buerger's disease.
* Venipuncture site located in area of insensitive skin; patients with a peripheral neuropathy including diabetic neuropathy.
* Patient intolerant of cold or with hypersensitivity to the cold.
* Patient unable or unwilling to give consent.
* Prior experience with vapocoolant spray
* Currently in another research trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon E. Mace, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farion KJ, Splinter KL, Newhook K, Gaboury I, Splinter WM. The effect of vapocoolant spray on pain due to intravenous cannulation in children: a randomized controlled trial. CMAJ. 2008 Jul 1;179(1):31-6. doi: 10.1503/cmaj.070874. PMID 18591524
- [Background] Hijazi R, Taylor D, Richardson J. Effect of topical alkane vapocoolant spray on pain with intravenous cannulation in patients in emergency departments: randomised double blind placebo controlled trial. BMJ. 2009 Feb 10;338:b215. doi: 10.1136/bmj.b215. PMID 19208703
- [Derived] Mace SE. Prospective, randomized, double-blind controlled trial comparing vapocoolant spray vs placebo spray in adults undergoing venipuncture. Am J Emerg Med. 2016 May;34(5):798-804. doi: 10.1016/j.ajem.2016.01.002. Epub 2016 Jan 7. PMID 26979261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: emergency department patients
Groups:
- Placebo (Normal Saline, Nature&Apos;s Tears): Application of sterile water stream (manufacturer above) for 4-10 seconds onto the venipuncture site.
  Sterile water (Nature's Tears): Topical stream of sterile water ( Nature's Tears ) 4-10 seconds duration to skin.
Period: Overall Study
Arm/Group | Placebo (Normal Saline, Nature&Apos;s Tears) | Vapocoolant (Pain Ease Medium Stream )
Started | 50 | 50
Completed | 50 (trial to enroll 50 in each group for total of 100) | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: pain after spray with placebo or vapocoolant
Groups:
- Nature's Tears: Application of sterile water stream (manufacturer above) for 4-10 seconds onto the venipuncture site.
  Sterile water (Nature's Tears): Topical stream of sterile water ( Nature's Tears ) 4-10 seconds duration to skin.
- Total: Total of all reporting groups
Arm/Group | Vapocoolant (Pain Ease Medium Stream ) | Nature's Tears | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.98 (13.42) | 51.48 (11.48) | 52.23 (12.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 23 | 54
  Male | 19 | 27 | 46
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Pain Scale on Numeric Rating Scale (NRS) ( 0 to 10)
Description: NRS scale: 0-10 ; No pain (0) - (5) moderate pain - Worst pain (10)
Time Frame: Less than 10 minutes after stream application.
Population: equal numbers in both groups by randomization to 50 in each group to look at NRS by change of 2 in NRS scale between the 2 groups
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vapocoolant (Pain Ease Medium Stream ) | Nature's Tears
Number analyzed (Participants) | 50 | 50
units on a scale | 1.7 (2.3) | 4.7 (2.9)

ADVERSE EVENTS:
Time Frame: 10 minutes
Description: Time frame = the time the patients were in the emergency department Skin assessments were done within 10 minutes after spray application
Arm/Group | Vapocoolant (Pain Ease Medium Stream ) | Nature's Tears
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 2/50 | 1/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vapocoolant (Pain Ease Medium Stream ) (N=50) | Nature's Tears (N=50)
Skin felt cool (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — "skin felt cool" at 10 minutes no skin abnormalities seen

LIMITATIONS AND CAVEATS:
This study enrolled only adults. No pediatric patients were enrolled. However, an earlier study by Farion KJ et al in CMAJ in 2008 found that the use of a vapocoolant (pain-ease) significantly decreased the pain of intravenous cannulation in children

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes